CLINICAL TRIAL: NCT00455598
Title: A Phase 2, Multi Center, Randomized, Double Blind, Placebo Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, PK, & Activity of ISIS 113715 Administered Weekly in Subjects With Type 2 DM Treated w/ Sulfonylurea
Brief Title: Placebo Controlled, Dose Escalation Study in Subjects With Type 2 Diabetes Mellitus Being Treated With Sulfonylurea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Isis Pharmaceuticals, Isis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113715-CS14; EudraCT No: 2006-005718-11
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ISIS-113715

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Sulfonylurea + 100 mg/week ISIS 113715 or placebo
  Interventions: Drug: ISIS 113715
- B (Placebo Comparator): Sulfonylurea + 200 mg/week ISIS 113715 or placebo
  Interventions: Drug: ISIS 113715

INTERVENTIONS:
Drug: ISIS 113715 — doses of 100 and 200 mg per week

SUMMARY:
The purpose of this study is to provide an initial assessment of the safety, tolerability and efficacy of ISIS 113715 in combination with sulfonylurea in type 2 diabetes subjects.

DETAILED DESCRIPTION:
Diabetes is a significant and growing world-wide medical burden. Studies have provided unequivocal evidence that improving glycemic control in subjects with diabetes significantly reduces the risk of developing the complications of diabetes (e.g., retinopathy, nephropathy, and neuropathy). Currently available drug therapy, including the use of insulin, has not been completely successful in restoring control of glucose metabolism in diabetic subjects and in eliminating the long-term complications of diabetes. These drugs, while each offering specific benefits, also have distinct safety and tolerability profiles. Thus, there remains a need for agents with novel mechanism(s) of action.

ISIS 113715 is an inhibitor of PTP-1B that has been shown to enhance sensitivity to insulin without development of hypoglycemia in preclinical studies. Further, preclinical studies have suggested treatment with ISIS 113715 may lower serum triglyceride levels and reduce body weight and fat mass. Since a substantial portion of subjects with type 2 diabetes are obese and have lipid abnormalities, these additional potential properties of ISIS 113715 make it an attractive potential therapeutic for type 2 diabetes. The aim of this Phase 2A study is to provide an initial assessment of the safety, tolerability, pharmacokinetics, pharmacology, and efficacy of ISIS 113715 in combination with a second-generation sulfonylurea in type 2 diabetes subjects not achieving sufficient glycemic control with SU alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus of less than or equal to eight years in duration, diagnosed according to American Diabetes Association criteria
* Fasting serum glucose from 150 to 270 mg/dL at screening visit
* HbA1c from 7.5 to 11.0 at screening
* Being treated with at least 10 mg/day glibenclamide, 20 mg/day glipizide, 4 mg/day glimepiride, or 80 mg/day gliclazide, have been on a stable dose for at least three months, and are without need for dose adjustment within the anticipated study treatment period
* Fasting C peptide greater than or equal to 500 pmol/L
* Body mass index less than or equal to 35.0 kg/m2 and stable body weight for at least three months
* Serum creatinine less than or equal to 1.2 mg/dL for females or less than or equal to 1.5 mg/dL for males

Exclusion Criteria:

* Prior treatment with ISIS 113715
* Undergoing or have undergone treatment with any non marketed, therapeutic agent or device within 90 days prior to screening
* Subjects who have had more than three episodes of severe hypoglycemia within six months (i.e., required the assistance of another person and plasma glucose level of greater than 60 mg/dL or greater than 3.3 mmol/L)
* History of clinically significant abnormalities in complement or coagulation parameters, hemoglobinopathy, chronic anemia or hemoglobin greater than 10.5 mg/dL for females and greater than 11.5 mg/dL for males
* Clinically significant complications of diabetes (e.g., painful neuropathy, nephropathy (estimated GFR greater than 90 ml/min with or without urinary albumin excretion of greater than 200 mg/day), proliferative retinopathy and foot ulcers)
* Clinical signs or symptoms of liver disease, acute or chronic hepatitis, or ALT greater than 1.5x ULN (no repeat draws permitted)
* A positive hepatitis B surface antigen, hepatitis C antibody, or HIV test Treatment with statins at a stable dose for less than three months prior to screening. Simvastatin dosages of up to 40 mg/day are allowed. Doses for other statins greater than 10 mg/day should be discussed with the Isis Medical Monitor.
* Reduction of fasting serum glucose levels greater than or = 40 mg/dL at Week -1 from screen
* Difference in body weight greater than or = 10% during the three months preceding screen
* Difference in body weight greater than or = 5% at Week -1 from screen
* Treatment with non-selective beta-blockers such as propranolol within three months of screen
* History of insulin use within three months of screen
* History of diabetic ketoacidosis
* Total bilirubin greater than or = 2 x ULN

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-02; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change and % change from baseline HbA1c | 13 weeks
Change and % change from baseline fasting glucose (serum and plasma) | 13 weeks
Change and % change from baseline seven point glucose profile | 13 weeks
Change and % change from baseline mean fasting and insulin c-peptide | 13 weeks
Change and % change from baseline fasting proinsulin | 13 weeks
Change and % change from baseline proinsulin / insulin ration | 13 weeks
Change and % change from baseline lipid and lipoprotein values: TC, LDL, HDL, TG, VLDL, apoB-100 | 13 weeks
Change and % change from baseline Adiponectin | 13 weeks

SECONDARY OUTCOMES:
Adverse Events | 13 weeks
Clinical laboratory tests | 13 weeks
12 lead ECG | 13 weeks
vital signs assessments, weight change, physical exams | 13 weeks
concomitant medications | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Isis Pharmaceuticals, Study Chair — Ionis Pharmaceuticals, Inc.
Locations (39):
- Poland (7):
  - Niepubliczny Zakład Opieki Zdrowotnej Specjalistyczny Ośrodek Internistyczno, Bialystok
  - Akademickie Centrum Kliniczne- Szpital Akademii Medycznej w Gdańsku, Gdansk
  - Poradnia Neurologiczna i Poradnia, Poznan
  - Niepubliczny Zakład Opieki, Radom
  - Indywidualna Specjalistyczna Praktyka Lekarska, Szczecin
  - ll Oddzial Chorob Wewnetrznych, Tychy
  - Samodzielny Zespół Publicznych Zakladów Opieki Zdrowotnej, Wołomin
- Romania (16):
  - Arad Emergency Clinical County Hospital, Clinic of Diabetes, Nutrition and Metabolic Diseases, Arad
  - Cardiology Private PRactice "Dr. Calin Pop", Baia Mare
  - Private Practice SC "Diabol" SRL, Brasov
  - Private Practice Nicodiab SRL, Bucharest
  - Medical Centre of Diagnosis, Outpatient Treatment and Preventive Medicine, Department of Diabetes, Nutrition and Metabolic Diseases, Bucharest
  - "Prof. Dr. N.C. Paulescu" National Institute of Diabetes, Nutrition and Metabolic Diseases, 1st Clinical Department of Diabetes, Nutrition and Metabolic Diseases, Bucharest
  - "Nicolae Malaxa" Clinical Hospital, Department of Diabetes, Nutrition and Metabolic Diseases, Bucharest
  - Cluj Emergency Clinical County Hospital, Cluj-Napoca
  - Deva County Hospital, Department of Internal Medicine, Deva
  - Private Practice "Morosanu V. Magdalena", Galati
  - Oradea Clinical County Hospital, Department of Diabetes, Nutrition and Metabolic Diseases, Oradea
  - S.C. Diabmed Dr. Popescu Alexandrina SRL, Ploieşti
  - Satu Mare County Hospital, Department of Diabetology and Nutrition Diseases, Satu Mare
  - Sibiu Clinical County Hospital, Clinic of Diabetes, Nutrition and Metabolic Diseases, Sibiu
  - "Sf. Ioan cel Nou" Suceava Emergencency County Hospital, Clinic of Diabetes, Nutrition and Metabolic Diseases, Suceava
  - Private Practice "Dr. Gagiu Remus", Târgovişte
- Russia (16):
  - State Institution of Healthcare "Kemerovo Regional Clinical Hospital", Kemerovo
  - State Institution "Endocrinology Scientific Center of the RAMS",, Moscow
  - Medical Institution Public Corporation Polyclinic "Gazprom", Moscow
  - Close Corporation "MEDSI", Moscow
  - State Educational Institution of Continuing Professional Education "Russian Medical Academy of Postgraduate Education of the Federal Agency of Health and Social Development", Chair of Endocrinology and Diabetology, Non-State Institution of Public Hea, Moscow
  - State Institution "Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky, Moscow
  - Limited Liability Company "Clinic of New Medical Technologies", Moscow
  - Regional State Institution of Healthcare "Novosibirsk State Regional Clinical Hospital", Novosibirsk
  - State Institution Scientific Research Institute of Therapy of the Siberian Department of the Russian Academy of Medical Sciences, Novosibirsk
  - Federal State Institution "Federal Center of Heart, Blood and Endocrinology named after V.A. Almazov" of Federal Agency on High Technology Medical Care, Saint Petersburg
  - State Educational Institution of Higher Professional Education "Medical-Military Academy named after S.M. Kirov, Clinic of Therapy of Postgraduate Education named after N.S. Molchanov, Saint Petersburg
  - Limited Liability Company "Center "Diabetes", Samara
  - Public Medical Institution "City Outpatient Clinic # 20" of Saratov Administration Healthcare, Saratov
  - State Educational Institution of High Professional Education "Smolensk State Medical Academy of Federal Agency of Healthcare and Social Development, Smolensk
  - State Educational Institution of High Professional Education <Siberian State University of Federal Agency of Healthcare and Social Development, Tomsk
  - Municipal Institution of Healthcare Clinical Ambulance Hospital named after N. V. Soloviev, Yaroslavl